CLINICAL TRIAL: NCT05884736
Title: Confirming the Permanent Cessation of Intracranial Circulation During Abdominal Normothermic Regional Perfusion After the Determination of Death by Circulatory Criteria
Brief Title: Confirming Permanent Lack of Blood Flow to the Brain During A-NRP DCC Organ Transplant
Acronym: CONCLUDE
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anton Skaro, Director of Liver Transplantation Surgery and Associate Professor - Department of Surgery, Western University, Canada
Other Study IDs: 4436
Record Dates: First submitted 2023-05-16; First posted 2023-06-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Organ Transplant
Keywords: A-NRP; neuromonitoring; brain activity; transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCC Donors: Standard criteria DCC donors will be undergoing the A-NRP perfusion process to recondition organs prior to procurement. Multimodal neuromonitors will be placed on the donor prior to withdrawal of life support and readings will be recorded during the withdrawal process and for the duration of the A-NRP perfusion process. The neuromonitoring team will be looking for evidence of brain blood flow or activity.
  Interventions: Other: Neuromonitoring

INTERVENTIONS:
Other: Neuromonitoring — Multimodal neuromonitoring will include: Transcranial colour-coded Doppler (TCCD), Electroencephalography (EEG), and Somatosensory evoked potentials (SSEP) or brainstem auditory evoked potentials (BAEP)

SUMMARY:
This study aims to evaluate the surgical technique used in Abdominal Normothermic Regional Perfusion (A-NRP) in death determination by circulatory criteria (DCC) organ donors. The proposed study will demonstrate that there is no resumption of brain blood flow or activity during the A-NRP procedure. This will be assessed using multimodal neuromonitoring protocol that enables continuous focused monitoring of brain blood flow and activity during A-NRP. This will provide evidence that brain blood flow and activity does not resume during NRP and ensure donor safety in using this technique in standard of care practice.

DETAILED DESCRIPTION:
This will be a multi-centre prospective observational cohort study that will enroll eligible DCC donors at participating donation hospitals. Participating programs will implement the A-NRP processes and organ recovery at the donation sites. Neurocritical care teams and donation physicians at the donation site and independent of transplant teams will implement neuromonitoring using the following modalities:

1. Transcranial colour-coded Doppler (TCCD) as a measure of brain blood flow,
2. Electroencephalography (EEG), as a measure of cortical brain electrophysiologic activity, and
3. Somatosensory evoked potentials (SSEP) or brainstem auditory evoked potentials (BAEP), as a measure of brainstem electrophysiologic activity.

The neuromonitoring team will interpret observed signals in real-time during the A-NRP process. This study will confirm whether current A-NRP surgical safeguards ensure maintenance of permanent cessation of brain blood flow and/or activity during A-NRP and will guide the adoption of A-NRP in Ontario.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 18 years of age
* Potential DCC donors whose families/surrogate decision makers have consented to DCC organ donation according to current criteria of the participating transplant programs. These may include patients donating a liver, kidneys, pancreas, and/or lungs; please see Appendix A for organ specific donor inclusion criteria.

Exclusion Criteria:

* < 18 years of age
* DCC donors who proceed to donation following medical assistance in dying or those who are able to provide first-person consent at the time of donation
* Injuries that anatomically preclude the use of neurological monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in critical care at participating study centers who qualify for DCC organ donation and whose families/surrogate decision makers have consented to DCC organ donation according to current criteria of the participating transplant programs.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Donor resumption of brain blood flow and/or activity | Through study completion, an average of 1 year
  Proportion of enrolled patients who have resumption of brain blood flow and/or activity during A-NRP on any neuromonitor and that is confirmed by neurocritical care physician and that results in termination of A-NRP

SECONDARY OUTCOMES:
Donor accrual rate | Through study completion, an average of 1 year
  Number of eligible donors who are enrolled in the study and complete study procedures
Consent rate | Through study completion, an average of 1 year
  Number of donors who consent to study procedures divided by the number of donors approached for study consent (target ≥ 80%)
Neuromonitoring modalities | Through study completion, an average of 1 year
  Number of neuromonitoring modalities used per patient and reasons for excluding specific modalities
Duration and proportion of neuromonitoring signal | Through study completion, an average of 1 year
  Duration of continuous neuromonitoring and proportion of total recording time with adequate signal per patient (velocity waveforms for TCCD, uv/mm for EEG, brainstem auditory evoked potentials (BAEP) signal, and somatosensory evoked potentials (SSEP) signal)
Neuromonitoring failure | Through study completion, an average of 1 year
  Proportion of enrolled patients who had failure of neuromonitoring equipment during recording

CONTACTS AND LOCATIONS:
Overall Officials: Anton Skaro, MD PhD, Principal Investigator — London Health Sciences Centre/Lawson Health Research Institute
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No